CLINICAL TRIAL: NCT01972061
Title: Foot/Hand Neuromodulation for Overactive Bladder (OAB)
Acronym: FootStim
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of continued funding
Sponsor: Christopher J Chermansky, MD (Other)
Responsible Party: Sponsor-Investigator, Christopher J Chermansky, MD, Assistant Professor of Urology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO13020474
Record Dates: First submitted 2013-10-18; First posted 2013-10-30 (Estimated); Results first posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CMG group (Experimental): Foot stimulation will be applied during a cystometrogram (CMG).
  Interventions: Device: Foot stimulation
- 3 hours group (Active Comparator): Foot stimulation will be applied daily for 3 hours in the evening.
  Interventions: Device: Foot stimulation
- 1/2 hour group (Active Comparator): Foot stimulation will be applied daily for 1/2 hour in the evening.
  Interventions: Device: Foot stimulation
- 3 hour hand group (Active Comparator): Hand stimulation will be applied daily for 3 hours in the evening.
  Interventions: Device: Foot stimulation

INTERVENTIONS:
Device: Foot stimulation — Foot stimulation electrically activates the somatic afferent nerves in the foot using FDA-approved, commercially available transcutaneous electrical nerve stimulator (TENS) and skin surface electrodes attached to the foot.

SUMMARY:
The purpose of this study is to determine if electrical stimulation of the foot is effective in the treatment of overactive bladder conditions.

DETAILED DESCRIPTION:
Foot neuromodulation is designed to treat OAB conditions by electrically stimulating the somatic afferent nerves in the foot using skin surface electrodes. The foot stimulation is non-invasive, can be performed at home, and has no adverse effects. Foot neuromodulation therapy will likely be accepted by more patients and have the potential to make a broader impact on the improvement of OAB conditions.

ELIGIBILITY:
Inclusion Criteria:

1. 18 year old men and women and older
2. Currently having overactive bladder (OAB) symptoms, i.e. urgency, frequency, or incontinence
3. No evidence of neurological disorder or urinary tract infection, i.e. clinically diagnosed as idiopathic OAB

Exclusion Criteria:

1. Pregnant women in their late pregnancy phase will be excluded because the increasing size of the baby/uterus may cause overactive bladder.
2. Patients with implanted electrical stimulators such as pacemaker will be excluded for potential interference with the TENS stimulator.
3. Patients who are allergic to Cipro or Bactrim will be excluded from the CMG study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-03; Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Chermansky, MD, Principal Investigator — University of Pittsburgh; Dawn McBride, RN, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CMG Group | 3 Hours Group | 1/2 Hour Group
Started | 1 | 23 | 20
Completed | 1 | 23 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The funding was not available to complete the 3 hour hand group.
Groups:
- Total: Total of all reporting groups
Arm/Group | CMG Group | 3 Hours Group | 1/2 Hour Group | Total
Number analyzed (Participants) | 1 | 23 | 20 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 11 | 11 | 22
  >=65 years | 1 | 12 | 9 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 23 | 20 | 44
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 23 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 0 | 20 | 19 | 39
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 23 | 20 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Urinary Incontinence Episodes Per Day
Description: Participants kept a daily voiding diary during week 1 (baseline), week 2 (foot stimulation), and week 3 (post foot stimulation). The average number per day urinary incontinence episodes was calculated for week 1 and week 2 for each subject.
Time Frame: Week 1, Week 2, Week 3
Measure: Mean (Standard Deviation); unit: Urinary Incontinence Episodes
Arm/Group | 3 Hours Group | 1/2 Hour Group
Number analyzed (Participants) | 23 | 20
Urinary Incontinence Episodes
  Week 1 | 3.7 (0.4) | 5.3 (0.4)
  Week 2 | 2.8 (0.4) | 4.3 (0.3)
  Week 3 | 2.8 (0.3) | 4.0 (0.3)

2. Secondary Outcome: Number of Urinary Urgency Episodes Per Day
Description: Participants kept a daily voiding diary during week 1 (baseline), week 2 (foot stimulation), and week 3 (post foot stimulation). The average number per day urinary urgency episodes was calculated for week 1 and week 2 for each subject.
Time Frame: Week 1, Week 2, Week 3
Measure: Mean (Standard Deviation); unit: Urinary urgency episodes per day
Arm/Group | 3 Hours Group | 1/2 Hour Group
Number analyzed (Participants) | 23 | 20
Urinary urgency episodes per day
  Week 1 | 7.6 (0.4) | 8.1 (0.3)
  Week 2 | 6.6 (0.3) | 8.0 (0.3)
  Week 3 | 6.6 (0.3) | 8.0 (0.3)

3. Other Pre Specified Outcome: Bladder Volume as Recorded on CMG for Strong Desire to Void
Description: Subject reports to the clinic for two CMGs. CMG #1 is the baseline measurement. CMG #2 is recorded during Foot Stimulation
Time Frame: CMG #1 and CMG#2
Measure: Number; unit: ml
Arm/Group | CMG Group
Number analyzed (Participants) | 1
ml
  CMG#1 Baseline | 265
  CMG #2 Foot Stimulation | 255

4. Other Pre Specified Outcome: Number of Urinary Voids Per Day
Description: Participants kept a daily voiding diary during week 1 (baseline), week 2 (foot stimulation) and week 3 (post foot stimulation)
Time Frame: Week 1, Week 2, Week 3
Measure: Mean (Standard Deviation); unit: urinary voids per day
Arm/Group | 3 Hours Group | 1/2 Hour Group
Number analyzed (Participants) | 23 | 20
urinary voids per day
  Week 1 | 9.1 (0.3) | 8.7 (0.3)
  Week 2 | 7.3 (0.3) | 8.5 (0.2)
  Week 3 | 7.3 (0.3) | 8.5 (0.2)

ADVERSE EVENTS:
Time Frame: 3 Weeks at the individual participant level.
Description: Adverse events were tracked from the time of consent until study completion. The study team followed the data safety and monitoring plan outlined in the protocol. The Principal Investigator and study team reviewed the data at regular intervals to assess, record and report any Adverse Events or Serious Adverse Events.
Arm/Group | CMG Group | 3 Hours Group | 1/2 Hour Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/23 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/1 | 0/23 | 0/20

LIMITATIONS AND CAVEATS:
The 3 hour hand group was not started or completed due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT01972061/Prot_SAP_000.pdf